CLINICAL TRIAL: NCT04945434
Title: Clinical Results of Chronic Cavitary Long-bone Osteomyelitis Treatment Using S53P4 Bioactive Glass; a Multi-center Study
Brief Title: Clinical Effectiveness of S53P4 Bioactive Glass in Treatment of Long-bone Chronic Osteomyelitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Tom van Vugt, Principal Investigator, Orthopedic Resident, Academisch Ziekenhuis Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUMC_METC174084
Record Dates: First submitted 2021-05-31; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Osteomyelitis; Bone Infection; Non-Union Fracture; Bone Infection of Lower Leg; Bone Infection of Pelvis, Hip, or Femur
Keywords: Bioactive glass; S53P4 BAG; Bonalive; Chronic Osteomyelitis
MeSH Terms: conditions — Osteomyelitis; Fractures, Ununited

STUDY DESIGN:
Intervention Model Description: Single group cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S53P4 BAG intervention group (Experimental): Patients recruited and enrolled in study for treatment with S53P4 BAG
  Interventions: Device: S53P4 bioactive glass (BonAlive)

INTERVENTIONS:
Device: S53P4 bioactive glass (BonAlive) — Surgical implantation of S53P4 in a bone defect created during debridement for chronic osteomyelitis.
  Other Names: Bonalive bioactive glass

SUMMARY:
This clinical trial studies the clinical effectiveness of S53P4 bioactive glass (BAG) as a bacterial growth inhibiting bone graft substitute in a one-stage or two-stage surgical procedure for treatment of chronic long bone osteomyelitis.

DETAILED DESCRIPTION:
In this prospective multicenter study, patients from two different university hospitals in the Netherlands were included. Treatment consisted of debridement surgery, implantation of S53P4-BAG, if necessary wound closure by a plastic surgeon and additional culture based systemic antibiotics. Primary outcome was eradication of infection based on clinical presentation, radiographic imaging and laboratory tests. Secondary analysis was performed on probable risk factors for treatment failure after S53P4-BAG implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical, radiographic and/or laboratory study confirmed chronic osteomyelitis of long bones
* Patients who are physically and mentally willing and able to comply with postoperative functional evaluation.
* Patients that can read and understand the Dutch language.

Exclusion Criteria:

* Patients with an diabetic ulcer related chronic osteomyelitis
* Patients that are pregnant.
* Patients who are unwilling to cooperate with the study protocol and follow-up schedule.
* Patients who, as judged by the surgeon, are mentally incompetent or are likely to be non-compliant with the prescribed post-operative routine and follow-up evaluation schedule.
* Patients with malignancy - active malignancy within last 1 year
* Patients known with a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the study (severe osteoporosis requiring medication, Paget's disease, renal osteodystrophy,hypercalcemia ) or is immunologically suppressed, or receiving steroids in excess of physiologic dose.
* Patients with a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
* Patients with systemic or metabolic disorders leading to progressive bone deterioration
* Patients with other concurrent illnesses that are likely to affect their outcome such as all autoimmune diseases (including RA), sickle cell anaemia, systemic lupus erythematosus, psoriasis, not controlled type 1/2 diabetes or renal disease requiring dialysis.
* Patients with a known sensitivity to device materials
* Patients that are an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Eradication of infection In clinical presentation | 1-5 years follow-up
  Based on the following Clinical Signs:
  - Absence of a draining fistula, redness, swelling, pain and fever (>38,5 degrees of celcius)
Absence of signs of chronic osteomyelitis on radiographic imaging (1/2) | 1 - 5 years follow-up
  Radiographic analysis of X-ray or CT images of the affected bone Based on a combination of 2 different infection paramaters
  Parameter 1:
  - Bone destruction
Absence of signs of chronic osteomyelitis on radiographic imaging (2/2) | 1 - 5 years follow-up
  Radiographic analysis of X-ray or CT images of the affected bone Based on a combination of 2 different infection paramaters
  Parameter 2:
  - Periostal reactions
Eradication of infection in blood sample analysis (1/3) | 1 - 5 years follow-up
  Based on a combination of 3 different infection parameters; parameter 1 is C-Reactive protein (<10mg/L), collected from a venapuncture.
Eradication of infection in blood sample analysis (2/3) | 1 - 5 years follow-up
  Based on a combination of 3 different infection parameters; parameter 2 is Leukocyte count (<11 x 10E9 cells/L); collected from a venapuncture.
Eradication of infection in blood sample analysis (3/3) | 1 - 5 years follow-up
  Based on a combination of 3 different infection parameters; parameter 3 is Erythrocyte Sedimantation Rate (<22mm/hour) collected from a venapuncture.

SECONDARY OUTCOMES:
Complication registration | 1-5 years follow-up
  Number of patients with adverse reactions or events related to S53P4 bioactive glass treatment

OTHER OUTCOMES:
Identification of possible risk factors for failure (1/10) | Pre-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 1:
  - Age at sugery (Years)
Identification of possible risk factors for failure (2/10) | Pre-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 2:
  - Gender (M/F)
Identification of possible risk factors for failure (3/10) | Pre-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 3:
  - BMI (kg/m2)
Identification of possible risk factors for failure (4/10) | 1-5 years follow-up
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 4:
  - Smoking (Yes/No)
Identification of possible risk factors for failure (5/10) | Pre-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 5:
  - Preoperative Cierny-Mader classification (1/2/3/4)
Identification of possible risk factors for failure (6/10) | Pre-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 6:
  - Presence of a preoperative fistula (number of patients)
Identification of possible risk factors for failure (7/10) | Postoperative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 7:
  - Mono- vs. Polybacterial peroperative culture (number of patients)
Identification of possible risk factors for failure (8/10) | Per-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 8:
  - One stage vs. Two stage surgical procedure (number of patients)
Identification of possible risk factors for failure (9/10) | Per-operative value (not time related)
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 9:
  - Closure of wound by a plastic surgeon (Yes/No)
Identification of possible risk factors for failure (10/10) | 1-5 years follow-up
  We identified a subset of 10 parameters that might be associated with the possible risk of failure of treatment and will be analyzed.
  Parameter 10:
  - Complications (number of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Arts, PhD, Study Chair — Maastricht Univeristy Medical Centre (MUMC+)